CLINICAL TRIAL: NCT05941364
Title: Factors Affecting the Sustainable Improvement of Nurses' Competency After Receiving an Evidence-based Practice Training Program
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Elhabashy, lecturer, Cairo University
Other Study IDs: NHTMRI-IRB 13-23
Record Dates: First submitted 2023-05-24; First posted 2023-07-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Evidence-based Practice
Keywords: Evidence-based Practice; Clinical Competency; Sustainability; Nurses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evidence-based practice (EBP) is a problem-solving and decision-making approach to improving the quality of care and closing the malpractice gap, especially for critical care nurses. Critical care nurses are responsible for the assessment of patients and the provision of care in intensive care units (ICUs). Critical care nurses need expertise and evidence to recognize clinical changes and prevent patient complications.

Despite the emphasis on EBP being applied in nurses' daily practice, a significant number of nurses have not gotten involved in EBP and are not fully aware of the concept of EBP. Nurses are unprepared to implement EBP due to a lack of information literacy skills in information searching and retrieval. Therefore, several studies have been conducted on the effects of different nursing skill training programs designed based on evidence. The almost short-term effect of the EBP training program is likely to be successful. Nevertheless, there is little evidence regarding the sustainability effects of these training activities over time. Therefore, the study aims to explore the factors affecting the sustainable improvement of nurses' competency after receiving an evidence-based practice training program.

Research question What are the factors that affect the sustainable improvement of nurses' competency after receiving an evidence-based practice training program? Study design A mixed, sequential method design with one qualitative and one quantitative method will be utilized in the study to facilitate a more comprehensive evaluation of the factors affecting the sustainable improvement of nurses' competency after receiving an EBP training program. We identified these factors from reviewing the literature

Study variables The study variables of this study are the factors affecting the sustainable improvement of nurses' competency after receiving an evidence-based practice training program. qualitative and quantitative research methods will be used, four main factors will be assessed quantitatively using the following four measurement adopted instruments.

-Sustained Implementation Support Scale (SISS)

Self-efficacy: General Self-Efficacy Scale (GSE):

Self-regulation: Self-Regulation Questionnaire (SRQ) The seven subscales

Motivation assessment scale:

The reliability and validity of the quantitative measuring tool content and face validity will be checked to ensure that the tools measure specifically what the study intends to measure. Internal consistency (Cronbach's alpha) will be used. Also, trustworthiness will be established for qualitative findings.

DETAILED DESCRIPTION:
Evidence-based practice (EBP) is a problem-solving and decision-making approach to improving the quality of care and closing the malpractice gap, especially for critical care nurses. Critical care nurses are responsible for the assessment of patients and the provision of care in intensive care units (ICUs). Critical care nurses need expertise and evidence to recognize clinical changes and prevent patient complications.

Despite the emphasis on EBP being applied in nurses' daily practice, a significant number of nurses have not gotten involved in EBP and are not fully aware of the concept of EBP. Nurses are unprepared to implement EBP due to a lack of information literacy skills in information searching and retrieval. Therefore, several studies have been conducted on the effects of different nursing skill training programs designed based on evidence. The almost short-term effect of the EBP training program is likely to be successful. Nevertheless, there is little evidence regarding the sustainability effects of these training activities over time. Therefore, the study aims to explore the factors affecting the sustainable improvement of nurses' competency after receiving an evidence-based practice training program.

Research question What are the factors that affect the sustainable improvement of nurses' competency after receiving an evidence-based practice training program? Study design A mixed, sequential method design with one qualitative and one quantitative method will be utilized in the study to facilitate a more comprehensive evaluation of the factors affecting the sustainable improvement of nurses' competency after receiving an EBP training program.

The inductive, category-generating qualitative approach will be employed using in-depth focus group semi-structured interview techniques to explore the participants' own experiences, beliefs, and perceptions using an open-ended question based on the participants' statements for addressing the contributing factors that affect the sustained implementation of the given EBPNTP into real-world practices. without the influence of supplementary texts or the researcher's internal suppositions.

Study variables The study variables of this study are the factors affecting the sustainable improvement of nurses' competency after receiving an evidence-based practice training program. qualitative and quantitative research methods will be used, four main factors will be assessed quantitatively using the following four measurement adopted instruments.

-Sustained Implementation Support Scale (SISS)

Self-efficacy: General Self-Efficacy Scale (GSE):

Self-regulation: Self-Regulation Questionnaire (SRQ) The seven subscales

Motivation assessment scale:

The reliability and validity of the quantitative measuring tool content and face validity will be checked to ensure that the tools measure specifically what the study intends to measure. Internal consistency (Cronbach's alpha) will be used. Also, trustworthiness will be established for qualitative findings.

Data collection procedure After obtaining the ethical approval of the IRB and the nurses' agreement to participate, the purpose and method of the research will be explained to nurses. the qualitative will start first by establishing a focus group interview based on predetermined interview guidelines. Then quantitative method will start by asking the nurses to respond to the self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* ICU nurses.
* nurses who took the EBP Training Program.

Exclusion Criteria:

- not willing to participate

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants sample and setting The study will be conducted in adult ICUs at the NHTMRI in Cairo, Egypt. The total capacity of the ICUs is 14 beds, divided into two sections. All nurses who participated as an intervention group (n = 37) in a previously unpublished yet study entitled "Effect of Evidence-Based Nursing Practices Training Program on the Competency of Nurses Caring for Mechanically Ventilated Patients: A Randomized Controlled Trial" who received the evidence-based nursing practice training program (EBNPTP) will be invited to participate in the current study.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
This is an observational study. Four questionnaires will be aggregated to assess one reported variable : The variable is (factor affecting the sustainable improvement of nurses' competency after receiving an EBP training program). | up to 3 weeks
  The four specific inventories are;
  1. Sustained Implementation Support Scale: 28-item measure assessing five categories of common barriers and enablers of sustained educational program implementation, 5-point scale from 1 (strongly disagree) to 5 (strongly agree).
  2. Self-efficacy Scale: 10 items used to measure how much people believe they can achieve their goals, despite difficulties, 4-point scale from 1 (Not at all true) to 4 (Exactly true).
  3. Self-regulation Questionnaire: 63 items, employed to measure the generalized ability to regulate behavior, 5-point scale from 1 (strongly disagree) to 5 (strongly agree).
  4. Motivation assessment scale: 12 items were used that correspond to intrinsic and extrinsic self-motivating factors, 5-point scale from 1 (strongly disagree) to 5 (strongly agree).
  The average item score will be used; the assessed factors with higher scores mean it has a higher contribution.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elhabashy S, Moriyama M, Saleh MA. Factors Affecting Sustainable Improvement of Nurses' EBP Competency After Receiving an EBP Training Program: A Mixed-Methods Study. J Clin Nurs. 2025 Sep 9. doi: 10.1111/jocn.70100. Online ahead of print. PMID 40922703